CLINICAL TRIAL: NCT06475404
Title: Open-label Multi-cohort Study of the Tolerability, Safety, and Pharmacokinetics of GNR-055 in Healthy Volunteers After a Single Intravenous Injection in Increasing Doses
Brief Title: A Study of the Tolerance, Safety, and Pharmacokinetics of GNR-055 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IDB-MPS-I02
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Mucopolysaccharidosis Type II; Metabolic Diseases
Keywords: Mucopolysaccharidosis type II; Mucopolysaccharidoses; Metabolic Diseases; Lysosomal Storage Diseases; Carbohydrate Metabolism; Inborn; Metabolism; Genetic Diseases; Neurobehavioral Manifestations; Neurologic Manifestations; Genetic Diseases, X-Linked
MeSH Terms: conditions — Mucopolysaccharidosis II; Metabolic Diseases; Mucopolysaccharidoses; Lysosomal Storage Diseases; Genetic Diseases, Inborn; Neurobehavioral Manifestations; Neurologic Manifestations; Genetic Diseases, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- verenafusp alfa 6 mg/kg intravenously (Experimental): Single intravenous administration
  Interventions: Biological: verenafusp alfa 6 mg/kg
- verenafusp alfa 9 mg/kg intravenously (Experimental): Single intravenous administration
  Interventions: Biological: verenafusp alfa 9 mg/kg
- verenafusp alfa 12 mg/kg intravenously (Experimental): Single intravenous administration
  Interventions: Biological: verenafusp alfa 12 mg/kg

INTERVENTIONS:
Biological: verenafusp alfa 6 mg/kg — Single intravenous administration of 6 mg/kg of verenafusp alfa
  Other Names: GNR-055
  Arms: verenafusp alfa 6 mg/kg intravenously
Biological: verenafusp alfa 9 mg/kg — Single intravenous administration of 9 mg/kg of verenafusp alfa
  Other Names: GNR-055
  Arms: verenafusp alfa 9 mg/kg intravenously
Biological: verenafusp alfa 12 mg/kg — Single intravenous administration of 12 mg/kg of verenafusp alfa
  Other Names: GNR-055
  Arms: verenafusp alfa 12 mg/kg intravenously

SUMMARY:
It is a phase I open-label single-dose, dose-escalation cohort study to evaluate of the tolerance, safety, and pharmacokinetics of GNR-055 in healthy volunteers

DETAILED DESCRIPTION:
GNR-055 (verenafusp alfa) is intended for enzyme replacement therapy (ERT) in patient with Mucopolysaccharidosis type II (MPS II), or Hunter syndrome. MPS II is a lysosomal storage disease with an X-linked recessive inheritance type, which is characterized by a decrease in the activity of the lysosomal enzyme iduronate-2-sulfatase (I2S), caused by a mutation in the idursulfase (IDS) gene. Enzyme deficiency leads to the accumulation of glycosaminoglycans (GAG) in lysosomes, mainly fractions of heparan and dermatan sulfates. Because of the insufficient activity of iduronate sulfatase participating in the first stage of catabolism of GAG, they accumulate in lysosomes of almost all types of cells of various tissues and organs. The disease is manifested by growth retardation, damage of many organs and systems, severe deformations of bones and joints, gross facial features, pathology of the respiratory and cardiovascular systems, damage to parenchymal organs (hepatosplenomegaly), hearing impairment. A severe form of the disease occurs with the involvement of the nervous system in the pathological process, including mental retardation, behavior anomalies, and impaired motor function.

GNR 055 (verenafusp alfa) is a modified enzyme I2S capable of penetrating the blood-brain barrier and thus it is expected to prevent neurodegenerative consequences and the development of cognitive deficit in the future that will allow achieving a significant improvement in the life quality and expectancy of patients with MPS II.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 45 years (inclusive) at the time of signing the Informed Consent Form;
* Body mass index (BMI) 18.5 to 29.9 kg/m2, body weight of 50 to 90 kg;
* A verified diagnosis as "healthy" (the diagnosis "healthy" is established based on a detailed medical history, in the absence of deviations from normal values during a clinical examination, including measurement of blood pressure, respiratory rate, heart rate, body temperature, laboratory and instrumental (ECG) examination data);
* A written informed consent to participate in the study in accordance with applicable laws in place and compliance with all the procedures and requirements/restrictions provided for by the study protocol;
* Consent to use adequate methods of contraception (double barrier method-male or female (for partners of male research volunteers), condom with spermicide, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, cervical cap with spermicide).

Exclusion Criteria:

* Known hypersensitivity to idursulfase and/or to the medicinal product excipients;
* Burdened allergy history;
* Drug intolerance;
* History of seizures;
* Deposit injections or implants use of any other medicinal product three months before the Screening Visit;
* An unusual way of living (night working, extreme physical activity);
* Diarrhea dehydration, vomiting, or other causes within 24 hours before the Screening Visit;
* Deviations from the normal values of the clinical, laboratory, and ECG examinations;
* If there are acute or chronic diseases of the cardiovascular, bronchopulmonary, nervous, immune, and endocrine systems, diseases of the gastrointestinal tract, liver and biliary tract, kidney and urinary tract, blood and lymphatic system, a history of mental illness;
* Positive results for hepatitis B or C markers, human immunodeficiency virus (HIV), and syphilis;
* Acute infectious diseases less than four weeks before the Screening Visit;
* Regular administration of medicinal products less than two weeks before the Screening Visit;
* Systolic blood pressure (SBP) below 90 mm Hg or above 139 mm Hg; diastolic blood pressure (DBP) below 50 mm Hg or above 89 mm Hg; heart rate (HR) below 60 bpm or above 90 bpm;
* Blood donation (450 mL or more of blood or plasma) less than three months before the Screening Visit;
* Participation in human clinical studies of medicinal products less than three months before the Screening Visit;
* Consumption of more than 5 units of alcohol per week (1 unit of alcohol is equal to 30 ml of ethyl alcohol) OR history of alcoholism, drug addiction, or drug abuse;
* Alcohol exhale positive test;
* Drug addiction and positive urine analysis for potent and narcotic substances;
* Smoking more than 5 cigarettes per day;
* Any planned surgical intervention during the study period;
* Reluctance to comply with contraceptive methods;
* Vaccination (with any vaccine) within 30 days before signing the informed consent and/or the need for vaccination during the study period; 23. History of an autoimmune disease; 24. History of any cancer.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As a rule, boys suffer from Mucopolysaccharidosis type II
Enrollment: 18 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with Adverse Events | Day 28
  Adverse events, Laboratory tests, Vital signs, Physical examination, 12-lead electrocardiogram, Allergic reactions, Infusion reactions, Antidrug antibody

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) | Day 4
  Analysis of equivalence of area under concentration-time curve from time 0 (predose) to the last quantifiable data point and to infinity
Pharmacokinetics: Peak Plasma Concentration (Cmax) | Day 4
  Analysis of equivalence of Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — JSC GENERIUM
Locations (1):
- State budgetary healthcare institution of the city of Moscow "City Clinic No. 2 of the Moscow Health Department", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No